CLINICAL TRIAL: NCT02591368
Title: MiniTightRope Suspensionplasty Compared With Ligamentous Reconstruction Tendon Interposition for the Treatment of Basilar Thumb Arthritis. A Randomized Clinical Trial
Brief Title: MiniTightRope Suspensionplasty Compared With LRTI for the Treatment of Basilar Thumb Arthritis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Orlando Health, Inc. (Other)
Responsible Party: Principal Investigator, Brett Lewellyn, Attending, Orlando Health, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15.035.03
Record Dates: First submitted 2015-10-26; First posted 2015-10-29 (Estimated); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Arthritis; Joint Diseases
MeSH Terms: conditions — Arthritis; Joint Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (3):
- Ligament reconstr. tendon interposition (Active Comparator): Ligament reconstruction, tendon interposition.
  Interventions: Procedure: Ligament reconstruction tendon interposition
- Mini Tight rope with one-suture (Active Comparator): Mini Tight rope with one suture
  Interventions: Procedure: Suspensionplasty with one-suture construct
- Mini Tight rope with two-suture (Active Comparator): Mini Tight rope with two sutures
  Interventions: Procedure: Suspensionplasty with two-suture construct

INTERVENTIONS:
Procedure: Ligament reconstruction tendon interposition — In this procedure the trapezium is removed and one of the patient's own tendons (or portion of the tendon), usually the flexor carpi radialis or abductor pollicis longus, is passed through a drill hole in the thumb metacarpal and is used to suspend the first metacarpal base.
  Arms: Ligament reconstr. tendon interposition
Procedure: Suspensionplasty with one-suture construct — In this procedure the trapezium is removed and an Arthrex mini tightrope system using Fiberwire suture is drilled across the first metacarpal to the second metacarpal and is used to suspend the first metacarpal base instead of a tendon.
  Arms: Mini Tight rope with one-suture
Procedure: Suspensionplasty with two-suture construct — In this procedure the trapezium is removed and two Arthrex mini tightrope systems using Fiberwire sutures are drilled across the first metacarpal to the second metacarpal and are used to suspend the first metacarpal base instead of a tendon.
  Arms: Mini Tight rope with two-suture

SUMMARY:
This prospective randomized trial aims to ascertain differences in outcome measures for the operative treatment of basilar thumb arthritis by comparing the two most common surgical treatments: LRTI and mini tightrope suspensionplasty. The Investigators will evaluate both subjective and objective data to determine if a particular surgical method offers more favorable outcomes.

DETAILED DESCRIPTION:
The study will be a prospective randomized-controlled trial comparing LRTI and mini tightrope suspensionplasty for the surgical treatment of basilar thumb arthritis. Patients meeting operative criteria who present to Level One Orthopaedics at Orlando Health will be consented for study participation. Subsequently, consented patients will be randomized into one of three treatment arms: LRTI, suspensionplasty with one-suture construct and suspensionplasty with two-suture construct. The patient will be blinded prior to the procedure; however, the performing surgeon will not be able to be blinded. The patient will become un-blinded postoperatively when the performing surgeon informs them which method was used. The investigators will then follow the patients for 5 years to assess the primary and secondary outcomes (see below) and analyze the data with an intention-to-treat method before publishing the conclusions. Follow-up visits will occur at two weeks, one month, three months, six months, one year, and five years. Outcome measures will incorporate subjective and objective measures and will include the SF-36 and Disabilities of Arm, Shoulder & Hand (DASH) questionnaires, pinch/grip strength, visual analog pain scale, patient satisfaction and postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* Radiographically diagnosed Stage II-IV basilar thumb arthritis as described by the Eaton and Littler classification system on either the right or left hand.

Exclusion Criteria:

* To have a history of prior surgical intervention for basilar thumb arthritis, trauma to the hand or wrist, or debilitating injury to the upper extremity.
* Patients under the age of 18 or with a history of a debilitating neurologic injury, either acute or chronic, to the upper extremity will be excluded.
* Patients that are non-operative candidates due to medical comorbidities will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Disabilities of Arm, Shoulder & Hand (DASH) questionnaire | An average of 5 years.
  30-item questionnaire designed to measure physical function and symptoms in people with musculoskeletal disorders of the upper extremity
SF-36 patient survey scores | On the follow-up visits
  Commonly accepted functional outcome scores used to evaluate patients post-operatively
Patient satisfaction surveys | An average of 5 years.
  Patient-reported experiences on care received
Pinch/grip strength | An average of 5 years.
  the measurable ability to exert pressure with the hand, fingers, or both. It is measured by having a patient forcefully squeeze, grip, or pinch dynamometers; results are expressed in either pounds or kilograms of pressure.

SECONDARY OUTCOMES:
Visual pain scale | An average of 5 years.
  Unidimensional measure of pain intensity anchored by scores of 0 ["no pain"] and 10 [worst pain imaginable] at its extremes.

CONTACTS AND LOCATIONS:
Overall Officials: Brett Lewellyn, MD, Principal Investigator — Orlando Health
Locations (1):
- Orlando Health, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Henderson EB, Smith EC, Pegley F, Blake DR. Intra-articular injections of 750 kD hyaluronan in the treatment of osteoarthritis: a randomised single centre double-blind placebo-controlled trial of 91 patients demonstrating lack of efficacy. Ann Rheum Dis. 1994 Aug;53(8):529-34. doi: 10.1136/ard.53.8.529. PMID 7944639
- [Background] Davis TR, Brady O, Dias JJ. Excision of the trapezium for osteoarthritis of the trapeziometacarpal joint: a study of the benefit of ligament reconstruction or tendon interposition. J Hand Surg Am. 2004 Nov;29(6):1069-77. doi: 10.1016/j.jhsa.2004.06.017. PMID 15576217
- [Background] Yao J, Lashgari D. Thumb basal joint: Utilizing new technology for the treatment of a common problem. J Hand Ther. 2014 Apr-Jun;27(2):127-32; quiz 133. doi: 10.1016/j.jht.2013.12.012. Epub 2014 Jan 3. PMID 24491585